CLINICAL TRIAL: NCT04314427
Title: Early Glycaemic Control in Type 2 Diabetes Patients After Bariatric Surgery
Brief Title: Early Glycaemic Control in Type 2 Diabetes Patients After Bariatric Surgery; ECODABS
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: University Hospital, Antwerp (Other); Universitair Ziekenhuis Brussel (Other); Karolinska Institutet (Other); Hospital San Carlos, Madrid (Other); University Hospital, Ghent (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Ville Wallenius, Ass.Prof., Sahlgrenska University Hospital
Other Study IDs: 016/12
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: Glycemic control
MeSH Terms: interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastric by-pass: Roux-en-Y gastric bypass (RYGB); the stomach is divided with staplers to create a small gastric pouch, while the jejunum is divided 30 to 50 cm distal to the ligament of Treitz. The distal limb is then anastomosed to the small gastric pouch and a jejunojejunostomy is performed 50 to 150 cm distal from the gastrojejunostomy.
  Interventions: Procedure: Roux-en-Y gastric bypass
- Sleeve gastrectomy: Sleeve gastrectomy reduces the stomach size by vertical stapling
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass
  Groups: Gastric by-pass
Procedure: Sleeve gastrectomy
  Groups: Sleeve gastrectomy

SUMMARY:
Describe and characterize the time-course for improvement in glucose control after bariatric surgery in obese patients with type 2 diabetes

Compare these changes in glycemic control after different techniques for bariatric surgery

DETAILED DESCRIPTION:
Obesity and its ensuing metabolic complications such as type 2 diabetes mellitus, are exponentially increasing worldwide. * * The most effective treatment for obesity is bariatric surgery. * Different bariatric procedures are available. In the 1960's, the Roux-en-Y gastric bypass (RYGB) was developed, in which the stomach is divided with staplers to create a small gastric pouch, while the jejunum is divided 30 to 50 cm distal to the ligament of Treitz. The distal limb is then anastomosed to the small gastric pouch and a jejunojejunostomy is performed 50 to 150 cm distal from the gastrojejunostomy. Sleeve gastrectomy on the other hand, reduces the stomach size by vertical stapling. In the 1990's, gastric banding was developed, reducing the volume of the stomach by annular banding. The amount of excess body weight reduction varies among the different techniques, with 60% to 70% reported for RYGB*, 55% for sleeve gastrectomy* and up to 65% for gastric banding*. Worldwide, it is estimated that a total of 344000 procedures were performed in 2008. Roux-en-Y gastric bypass was the most common (47%) followed by gastric banding (42%) and sleeve gastrectomy (5%).*

In 1987, Pories et al. published data on the stunning observation that 99% of obese patients with type 2 diabetes or impaired glucose tolerance that had undergone Roux-en-Y gastric bypass became and remained euglycemic after surgery.* Since then, all commonly used bariatric procedures have been shown to restore a normal glucose profile in many diabetes patients. Current data suggest that the bypass procedures are more effective in doing so, with success rates up to 80%,* than the purely restrictive procedures such as sleeve gastrectomy and gastric banding, with success rates varying between 30% and 70%.* The improvement in glycaemic control is already seen a few days after surgery, long before any substantial weight loss occurs.

Although different reasons for the rapid amelioration in glycaemic control are discussed in literature, the exact underlying mechanisms are still not understood. In the restrictive procedures, the effect is thought to be mainly mediated by caloric restriction and the ensuing reduction in body weight and improvement in insulin resistance.* The malabsorptive procedures, such as RYGB, offer different explanatory possibilities. In the so-called 'fore-gut hypothesis', it is suggested that the exclusion of the duodenum and proximal jejunum may reduce insulin resistance. * The 'hind-gut hypothesis' on the other hand, suggests that it is the altered delivery of nutrients to the distal small bowel that causes exaggerated responses of the gut hormones. These gut hormones act as anorectic agents and as incretins that stimulate the beta cells in the pancreas to restore normal first phase insulin response. *

Most studies to investigate the alterations in glucose metabolism are performed weeks to months after surgery. There are limited data on the evolution of blood glucose in the first days and weeks after RYGB.* However, to our knowledge, no such data exist on the glycaemic control immediately after sleeve gastrectomy and gastric banding. With the present study we document the evolution in glycaemic control immediately after RYGB, sleeve gastrectomy and gastric banding in type 2 diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female type 2 diabetic patients
* Patients aged 18-65 years
* Diabetes treatment consisting of dietary measures or any of the following:
* Metformin
* Sulfonylurea
* Glinides
* Glitazones
* Acarbose
* Any type of insulin
* BMI ≥ 35 kg/m2

Exclusion Criteria:

* Active alcohol abuse
* Active psychiatric illness
* MODY (maturity onset diabetes of the young)
* Type 1 diabetes
* Diabetes treatment consisting of DPP IV-inhibitors or incretin mimetics
* Pregnancy and gestational diabetes
* Prior bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetes mellitus typ 2 and obesity
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Glucose control | from day one to 2-3 weeks after surgery
  the aim is to describe and characterize the time-course for improvement in glucose control after bariatric surgery in obese patients with type 2 diabetes

SECONDARY OUTCOMES:
Changes in glycemic control | day one post op to 2-3 weeks after surgery
  To compare these changes in glycemic control after different techniques for bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ville Wallenius, Ass. Prof., Principal Investigator — Sahlgrenska University Hospital
Locations (7):
- Belgium (3):
  - Antwerp University Hospital, Antwerp, Edegem
  - Universitair Ziekenhuis, Brussels, Jette
  - Gent University Hospital, Ghent
- Hospital Clinico San Carlos, Madrid, Spain
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska Institutet, Stockholm
- South kensington campus, London, United Kingdom